CLINICAL TRIAL: NCT02686918
Title: Feasibility Assessment of a Patients Follow-up Visit Receiving Trastuzumab Subcutaneous by Advanced Practice Nurse - TIPA
Brief Title: Feasibility Assessment of a Patients Follow-up Visit Receiving Trastuzumab Subcutaneous by Advanced Practice Nurse
Acronym: TIPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-01
Record Dates: First submitted 2016-02-08; First posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- consultation by Advanced Practice Nurse. (Experimental): During consultations, patients will be seen successively by Advanced Practice Nurse and referent oncologist.
  Interventions: Other: Advanced Practice Nurse consultation

INTERVENTIONS:
Other: Advanced Practice Nurse consultation

SUMMARY:
The main of this study is to assess the feasibility of a patients follow-up visit receiving trastuzumab subcutaneous by Advanced Practice Nurse.

ELIGIBILITY:
Inclusion Criteria:

* Patient care at the Cancer Institute Lucien Neuwirth
* Patient aged over 18 years
* Patient with breast cancer overexpressing HER2 adjuvant
* Patient having finished their chemotherapy treatment with IV followed the oncologist day hospital
* Patient under Trastzumab subcutaneously
* Patient affiliated or entitled to a social security scheme (mandatory requirement for all studies)

Exclusion Criteria:

* Refusal to participate, most patient protected under guardianship.
* Patient in inability to understand the course of the study
* Patient with documented history of cognitive or psychiatric disorders.
* Patients pregnant or lactating
* Patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of consultation requiring a medical advice between IPA and oncologist | 1 year
  Estimate the correlation between the IPA and the oncologist about whether or not a medical opinion during the consultation

SECONDARY OUTCOMES:
Percentage of consultations delegated to the IPA | 1 year
  The oncologist estimate the percentage of consultations can be delegated to the IPA
Physician satisfaction questionnaire | 1 year
  Physician satisfaction questionnaire of the delegation of his consultations to the IPA